CLINICAL TRIAL: NCT01024452
Title: Randomized Comparison of Warfarin Dosing Quality Between the Hamilton Nomogram and a Commercial Computer System
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Dr. S. Connolly, Population Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-283
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2009-12

CONDITIONS: Patients at Risk for Thrombosis
Keywords: anticoagulation; warfarin; computer systems; international normalized ratio; nomograms
MeSH Terms: interventions — Nomograms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- DAWN AC (Experimental)
  Interventions: Device: DAWN AC
- Hamilton Nomogram (Active Comparator)
  Interventions: Device: Hamilton Nomogram

INTERVENTIONS:
Device: DAWN AC — computerized dosing management system for anticoagulation clinics
  Other Names: DAWN AC, 4S Information Systems Ltd.
  Arms: DAWN AC
Device: Hamilton Nomogram — simple nomogram for warfarin maintenance dosing
  Other Names: Nomogram (algorithm)
  Arms: Hamilton Nomogram

SUMMARY:
Randomized comparison of warfarin dosing quality between the Hamilton nomogram and a commercial computer system.

Hypothesis: Mean TTR of patients managed with the commercial computer system is non-inferior to management with the validated Hamilton Nomogram.

DETAILED DESCRIPTION:
Warfarin has a variable effect and many potential food and drug interactions. To have an optimal therapeutic effect the International Normalized Ratio (INR) needs to be maintained within the therapeutic target range. The time that a patient spends within the therapeutic target range is an intermediate quality indicator for patient outcomes and should be optimized. For this purpose, we use in our anticoagulation clinic the simple two-step Hamilton nomogram, which has been validated by Kim et al. who showed that the nomogram improved INR control for warfarin maintenance compared with expertise-based dosing in our anticoagulation clinic (see references). Computer systems are also known to outperform expertise-based dosing, but no direct comparison of a computer system with a simple nomogram has been assessed. In this single-center randomized controlled clinical trial we will compare the simple two-step Hamilton nomogram with the widely used computerized dosing management system DAWN AC regarding their effect on time in therapeutic range for patients on maintenance dosing with target range 2-3.

ELIGIBILITY:
Inclusion Criteria:

* On warfarin maintenance therapy
* INR target range 2-3
* At least 3 historical INRs on maintenance therapy
* At least 1 historical INR in the last 3 months

Exclusion Criteria:

* Participation in another study
* On multiple pill strengths

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1298 (Actual)
Dates: Start 2009-11; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
TTR: The proportion of time a patient spends in the therapeutic INR range (2-3) | TTR calculated over the entire study period (6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Connolly, MD, Principal Investigator — Director, Division of Cardiology
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Poller L, Keown M, Ibrahim S, Lowe G, Moia M, Turpie AG, Roberts C, van den Besselaar AM, van der Meer FJ, Tripodi A, Palareti G, Shiach C, Bryan S, Samama M, Burgess-Wilson M, Heagerty A, Maccallum P, Wright D, Jespersen J; European Action on Anticoagulation (EAA). A multicentre randomised assessment of the DAWN AC computer-assisted oral anticoagulant dosage program. Thromb Haemost. 2009 Mar;101(3):487-94. PMID 19277410
- [Background] Kim YK, Nieuwlaat R, Connolly SJ, Schulman S, Meijer K, Raju N, Kaatz S, Eikelboom JW. Effect of a simple two-step warfarin dosing algorithm on anticoagulant control as measured by time in therapeutic range: a pilot study. J Thromb Haemost. 2010 Jan;8(1):101-6. doi: 10.1111/j.1538-7836.2009.03652.x. Epub 2009 Oct 14. PMID 19840361